CLINICAL TRIAL: NCT01576718
Title: A 12-Week Dose-ranging Study to Evaluate the Efficacy and Safety of Fp Spiromax® (Fluticasone Propionate Inhalation Powder) Administered Twice Daily Compared With Placebo in Adolescent and Adult Subjects With Severe Persistent Asthma Uncontrolled on High Dose Inhaled Corticosteroid Therapy
Brief Title: A Study of the Effectiveness and Safety of Different Doses of Fluticasone Propionate Taken From a Dry Powder Inhaler (Puffer) in Adolescents and Adults Who Have Asthma That is Not Controlled by High Dose Inhaled Corticosteroid Asthma Medications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FpS-AS-202; 2010-023601-35 (EudraCT Number)
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Asthma
Keywords: Dose ranging; Fluticasone Propionate; Dry Powder Inhaler (DPI); High Dose ICS; Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Fp MDPI 50 mcg (Experimental): Fluticasone propionate (Fp) 50 mcg per dose twice a day (for a total daily dose of 100 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol
- Fp MDPI 100 mcg (Experimental): Fluticasone propionate (Fp) 100 mcg per dose twice a day (for a total daily dose of 200 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol
- Fp MDPI 200 mcg (Experimental): Fluticasone propionate (Fp) 200 mcg per dose twice a day (for a total daily dose of 400 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol
- Fp MDPI 400 mcg (Experimental): Fluticasone propionate (Fp) 400 mcg per dose twice a day (for a total daily dose of 800 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol
- Placebo MDPI (Placebo Comparator): Placebo twice a day using a multidose dry powder inhaler (MDPI) for 12 weeks in a double-blind manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Other: Placebo MDPI; Drug: albuterol/salbutamol
- Flovent Diskus 250mcg (Active Comparator): Fluticasone propionate (Fp) 250 mcg per dose twice a day (for a total daily dose of 500 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in an open-label manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
  Interventions: Drug: Flovent Diskus; Drug: albuterol/salbutamol

INTERVENTIONS:
Drug: Fp MDPI — Fp MDPI is an inhalation-driven multidose dry powder inhaler (MDPI) containing fluticasone propionate (Fp) dispersed in a lactose monohydrate excipient and contained within a reservoir. A metered dose of drug is delivered to a dose cup via an air pulse activated when the cap is opened.
  During the treatment period, participants were randomized to 50, 100, 200 or 400 mcg of Fp one inhalation twice a day for a total daily dose of 100, 200, 400 or 800 mcg. Study drug was administered in the morning and in the evening.
  Other Names: fluticasone propionate; Fp SPIROMAX® Inhalation Powder
  Arms: Fp MDPI 100 mcg; Fp MDPI 200 mcg; Fp MDPI 400 mcg; Fp MDPI 50 mcg
Other: Placebo MDPI — Placebo multidose dry powder inhaler (MDPI) in the morning and evening. Placebo MDPI was provided in devices identical in appearance to Fp MDPI.
  Arms: Placebo MDPI
Drug: Flovent Diskus — Flovent Diskus contains the active ingredient fluticasone propionate (Fp). Flovent Diskus 250 mcg was used twice a day, once in the morning and evening, for a total daily dose of 500 mcg of Fp. This therapy was not blinded as the inhaler device was different than the MDPI used in the other treatment arms.
  Other Names: Fluticasone propionate
  Arms: Flovent Diskus 250mcg
Drug: albuterol/salbutamol — A short-acting β2-adrenergic agonists (SABA), albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI), was provided to be used as needed for the relief of asthma symptoms during both the run-in and treatment periods (to replace the subject's current rescue medication).
  Other Names: short-acting β2-adrenergic agonists

SUMMARY:
The primary objective of this study is to evaluate the dose response, efficacy and safety of 4 different doses of fluticasone propionate (50, 100, 200, and 400mcg) delivered as Fluticasone Spiromax® Inhalation Powder (Fp Spiromax) when administered twice daily in subjects 12 years of age and older with severe persistent asthma who are uncontrolled on high dose ICS therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent signed and dated by the subject and/or parent /legal guardian before conducting any study related procedure.
2. Male or female 12 years and older, as of the Screening Visit. Male or female 18 years and older, as of the Screening Visit, in countries where local regulations or the regulatory status of study medication permit enrollment of adults only.
3. General good health, and free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the subject at increased risk during the study.
4. Asthma Diagnosis: Asthma as defined by the National Institutes of Health (NIH).
5. Severity of Disease:

   • A best forced expiratory volume in one second (FEV1) of 40%-85% of the predicted normal value during the Screening Visit. NHANES III predicted values will be used for subjects aged ≥12 years and adjustments to predicted values will be made for African American subjects. ATS/ERS 2005 criteria for acceptability, reproducibility, and end of test must be met for spirometry
6. Reversibility of Disease: Demonstrated a ≥12% reversibility of FEV1 within 30 minutes following 2 inhalations of albuterol/salbutamol inhalation aerosol (if required, spacers are permitted for reversibility testing only) at the Screening Visit. If a subject fails to demonstrate an increase in FEV1 ≥12% then the subject is not eligible for the study and will not be allowed to re-screen. Reversibility values of 11.50 - 11.99 will be rounded to 12. Documented historical reversibility of ≥ 12 % within 3 months of the Screening Visit will be accepted.
7. Current Asthma Therapy: Subjects will be required to be on a short acting β2 agonist and inhaled corticosteroid for a minimum of 8 weeks before the Screening Visit and have been maintained on a stable dose of inhaled corticosteroids for four weeks prior to the Screening Visit at one of the following doses:

   * Fluticasone propionate HFA MDI ≥ 880 mcg/day
   * Fluticasone propionate DPI≥ 1000 mcg/day
   * Beclomethasone dipropionate DPI ≥ 2000 mcg/day
   * Beclomethasone dipropionate HFA (QVAR)≥ 640 mcg/day
   * Beclomethasone dipropionate HFA (Clenil Modulite)≥ 2000 mcg/day
   * Budesonide DPI ≥ 1600 mcg/day
   * Budesonide MDI ≥ 1600 mcg/day
   * Flunisolide ≥ 2000 mcg/day
   * Triamcinolone acetonide ≥ 2000 mcg /day
   * Mometasone furoate DPI ≥ 880 mcg/day
   * Ciclesonide HFA MDI ≥ 640 mcg/day

   Exception 1: Based upon the investigator's judgment that there is no inherent harm in changing the subject's current ICS/LABA therapy and the subject provides consent, subjects on inhaled Fluticasone propionate/salmeterol DPI ≥ 1000 mcg/day, or Fluticasone propionate/salmeterol HFA ≥ 880 mcg/day, or Fluticasone propionate/Formoterol ≥ 1000 mcg/day,or Beclomethasone dipropionate/Formoterol ≥ 400 mcg/day, or Budesonide/formoterol HFA ≥ 640 mcg/day, or Budesonide/formoterol DPI ≥ 800 mcg/day, or Mometasone furoate/formoterol MDI ≥ 800 mcg/day or subjects on a qualifying ICS dose plus a long-acting β2-agonists (LABA) administered via separate inhalers, may be switched to a qualifying dose of fluticasone propionate provided the subjects will not participate in the PK portion of the study.

   Exception 2: Subjects on a qualifying dose of fluticasone propionate who wish to participate in the PK portion of the study and who provide consent may have their fluticasone propionate switched to a different qualifying ICS (non-fluticasone propionate) at a pre-screening visit. The subject will be required to return to the clinic to complete the Screening Visit following a 1-week washout period.
8. Short-Acting β2-Agonists: All subjects must be able to replace their current short-acting β2-agonists with albuterol/salbutamol inhalation aerosol at the Screening Visit for use as needed for the duration of the study. The use of spacer devices with the metered dose inhaler (MDI) will not be allowed during the study with exception of it's use during reversibility testing at the Screening Visit. Nebulized albuterol/salbutamol will not be allowed at any time during the study. Subjects must be able to withhold all inhaled short-acting β2 sympathomimetic bronchodilators for at least 6 hours prior to all study visits.
9. If female, is currently not pregnant, breast feeding, or attempting to become pregnant, has a negative serum pregnancy test, and is of

   * Non-childbearing potential, defined as:

     * Before menarche, or
     * 1 year post-menopausal, or
     * Surgically sterile (tubal ligation, bilateral oophorectomy, or hysterectomy), or
     * Congenital sterility, or
     * Diagnosed as infertile and not undergoing treatment to reverse infertility or is of
   * Child-bearing potential, willing to commit to using a consistent and acceptable method of birth control as defined below for the duration of the study:

     * Systemic contraception used for 1 month prior to screening, including birth control pills, transdermal patch (Ortho Evra®), vaginal ring (NuvaRing®), levonorgesterel (Norplant®), or injectable progesterone (Depo-Provera®), or
     * Double barrier methods (condoms, cervical cap, diaphragm, and vaginal contraceptive film with spermicide), or
     * Intrauterine device (IUD) or
     * Monogamous with a vasectomized male partner or is of
   * Child-bearing potential and not sexually active, willing to commit to using a consistent and acceptable method of birth control as defined above for the duration of the study, in the event the subject becomes sexually active
10. Capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent/assent and being compliant with all study requirements (visits, record-keeping, etc).

Exclusion Criteria:

1. History of life-threatening asthma that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures.
2. Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that is not resolved within 2 weeks of the Screening Visit. In addition, the subject must be excluded if such infection occurs between the Screening Visit and the Randomization Visit.
3. Any asthma exacerbation requiring oral corticosteroids within 1 month of the Screening Visit. A subject must not have had any hospitalization for asthma within 2 month prior to the Screening Visit.

   Note: An exacerbation of asthma is defined as any worsening of asthma requiring any treatment other than rescue albuterol/salbutamol HFA MDI and/or the subject's regular inhaled corticosteroid maintenance treatment. This includes requiring the use of systemic corticosteroids and/or emergency room visit or hospitalization, a change in the subject's regular inhaled corticosteroid maintenance treatment, or the addition of other asthma medications.
4. Presence of glaucoma, cataracts, ocular herpes simplex, or malignancy other than basal cell carcinoma.
5. Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular (e.g., congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia or coronary heart disease), hepatic, renal, hematological, neuropsychological, endocrine (e.g., uncontrolled diabetes mellitus, uncontrolled thyroid disorder, Addison's disease, Cushing's syndrome), gastrointestinal (e.g., poorly-controlled peptic ulcer, GERD), or pulmonary (e.g., chronic bronchitis, emphysema, bronchiectasis with the need for treatment, cystic fibrosis, bronchopulmonary dysplasia, chronic obstructive pulmonary disease). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which could affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
6. Have any of the following conditions that, in the judgment of the investigator, might cause participation in this study to be detrimental to the subject, including, but not limited to:

   * Current malignancy excluding basal cell carcinoma; History of malignancy is acceptable only if the subject has been in remission for one year prior to the Screening Visit. (Remission is defined as no current evidence of malignancy and no treatment for the malignancy in the 12 months prior to the Screening Visit)
   * Current or untreated tuberculosis; History of tuberculosis is acceptable only if a subject has received an approved prophylactic treatment regimen or an approved active treatment regimen and has had no evidence of active disease for a minimum of 2 years
   * Uncontrolled hypertension (systolic BP ≥160 or diastolic BP >100)
   * Stroke within 3 months prior to the Screening Visit
   * Immunologic compromise
7. History of a positive test for HIV, hepatitis B or hepatitis C infection.
8. Untreated oral candidiasis at the Screening Visit. Subjects with clinical visual evidence of oral candidiasis and who agree to receive treatment and comply with appropriate medical monitoring may enter the study
9. History of any adverse reaction to any intranasal, inhaled or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the dry powder inhalers (Spiromax or Diskus) used in the study (i.e., lactose).
10. History of severe allergy to milk protein.
11. Use of systemic, oral or depot corticosteroids within 4 weeks prior to the Screening Visit

    * Use of topical corticosteroids (≤1% hydrocortisone cream) for dermatological disease is permitted
    * Use of intranasal corticosteroids or ocular corticosteroids at a stable dose for at least 4 weeks prior to the Screening Visit and throughout the study is permitted
12. Use of immunosuppressive medications within 4 weeks prior to the Screening Visit and during the study.
13. Immunotherapy for the treatment of allergy at a stable maintenance dose for at least 90 days prior to the Screening Visit and which will remain at a stable dose without escalation throughout the study is permitted.
14. Use of Cytochrome P450 3A4 (CYP3A4) inhibitors (e.g., ritonavir, ketoconazole, itraconazole) within 4 weeks prior to the Screening Visit. Strong and moderate CYP3A4 inhibitors are prohibited and weak CYP3A4 are allowed.
15. History of alcohol or drug abuse within two years preceding the Screening Visit.
16. Current smoker or a smoking history of 10 pack years or more (a pack year is defined as smoking 1 pack of cigarettes/day for 1 year). A subject may not have used tobacco products within the past one year (e.g., cigarettes, cigars, chewing tobacco, or pipe tobacco).
17. Study participation by clinical investigator site employees and/or their immediate relatives.
18. Study participation by more than one subject from the same household at the same time. However, after the study completion or discontinuation by one subject another subject from the same household may be screened.
19. Participation in any investigational drug study within the 30 days (starting at the final follow-up visit) preceding the Screening Visit or planned participation in another investigational drug study at any time during this study.
20. Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the subject's last study related visit (for eligible subjects only - if applicable). Eligible female subjects unwilling to employ appropriate contraceptive measures to ensure that pregnancy will not occur during the study will be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (300):
- United States (148):
  - Teva Investigational Site 10504, Birmingham, Alabama
  - Teva Investigational Site 10565, Homewood, Alabama
  - Teva Investigational Site 11527, Goodyear, Arizona
  - Teva Investigational Site 10516, Tucson, Arizona
  - Teva Investigational Site 10573, Bakersfield, California
  - Teva Investigational Site 11518, Costa Mesa, California
  - Teva Investigational Site 10590, Fountain Valley, California
  - Teva Investigational Site 10551, Granada Hills, California
  - Teva Investigational Site 11520, Huntington Beach, California
  - Teva Investigational Site 11545, Huntington Beach, California
  - Teva Investigational Site 10547, Long Beach, California
  - Teva Investigational Site 11549, Los Angeles, California
  - Teva Investigational Site 10503, Mission Viejo, California
  - Teva Investigational Site 10536, Newport Beach, California
  - Teva Investigational Site 10540, Orange, California
  - Teva Investigational Site 11551, Orange, California
  - Teva Investigational Site 10578, Palmdale, California
  - Teva Investigational Site 10585, Redwood City, California
  - Teva Investigational Site 11538, Rolling Hills Estates, California
  - Teva Investigational Site 11522, Roseville, California
  - Teva Investigational Site 10582, San Diego, California
  - Teva Investigational Site 11554, San Diego, California
  - Teva Investigational Site 10563, San Jose, California
  - Teva Investigational Site 11556, Santa Monica, California
  - Teva Investigational Site 10506, Stockton, California
  - Teva Investigational Site 10529, Walnut Creek, California
  - Teva Investigational Site 10545, Centennial, Colorado
  - Teva Investigational Site 10572, Colorado Springs, Colorado
  - Teva Investigational Site 10533, Denver, Colorado
  - Teva Investigational Site 11531, Denver, Colorado
  - Teva Investigational Site 11542, Denver, Colorado
  - Teva Investigational Site 11569, Wheat Ridge, Colorado
  - Teva Investigational Site 10528, Waterbury, Connecticut
  - Teva Investigational Site 10556, Boynton Beach, Florida
  - Teva Investigational Site 11513, Brandon, Florida
  - Teva Investigational Site 11507, Clearwater, Florida
  - Teva Investigational Site 11546, Fort Myers, Florida
  - Teva Investigational Site 11526, Hialeah, Florida
  - Teva Investigational Site 11525, Kissimmee, Florida
  - Teva Investigational Site 10537, Miami, Florida
  - Teva Investigational Site 10553, Miami, Florida
  - Teva Investigational Site 11508, Miami, Florida
  - Teva Investigational Site 11514, Miami, Florida
  - Teva Investigational Site 11516, Miami, Florida
  - Teva Investigational Site 11530, Miami, Florida
  - Teva Investigational Site 11570, Miami, Florida
  - Teva Investigational Site 10571, Ocala, Florida
  - Teva Investigational Site 11537, Sarasota, Florida
  - Teva Investigational Site 10593, South Miami, Florida
  - Teva Investigational Site 11555, Tallahassee, Florida
  - Teva Investigational Site 10554, Tamarac, Florida
  - Teva Investigational Site 10539, Tampa, Florida
  - Teva Investigational Site 10525, Valrico, Florida
  - Teva Investigational Site 11504, Albany, Georgia
  - Teva Investigational Site 10511, Columbus, Georgia
  - Teva Investigational Site 11510, Columbus, Georgia
  - Teva Investigational Site 11572, Columbus, Georgia
  - Teva Investigational Site 10568, Lawrenceville, Georgia
  - Teva Investigational Site 10586, Lilburn, Georgia
  - Teva Investigational Site 11539, Savannah, Georgia
  - Teva Investigational Site 10543, Stockbridge, Georgia
  - Teva Investigational Site 11558, Indianapolis, Indiana
  - Teva Investigational Site 10527, South Bend, Indiana
  - Teva Investigational Site 10584, Iowa City, Iowa
  - Teva Investigational Site 11501, Overland Park, Kansas
  - Teva Investigational Site 10591, Lexington, Kentucky
  - Teva Investigational Site 11567, Louisville, Kentucky
  - Teva Investigational Site 10513, Metairie, Louisiana
  - Teva Investigational Site 10564, Bangor, Maine
  - Teva Investigational Site 11548, Baltimore, Maryland
  - Teva Investigational Site 10510, Largo, Maryland
  - Teva Investigational Site 10577, Wheaton, Maryland
  - Teva Investigational Site 10538, Brockton, Massachusetts
  - Teva Investigational Site 10546, North Dartmouth, Massachusetts
  - Teva Investigational Site 11502, Troy, Michigan
  - Teva Investigational Site 10531, Plymouth, Minnesota
  - Teva Investigational Site 11562, Columbia, Missouri
  - Teva Investigational Site 11563, Columbia, Missouri
  - Teva Investigational Site 10552, St Louis, Missouri
  - Teva Investigational Site 10575, St Louis, Missouri
  - Teva Investigational Site 10589, St Louis, Missouri
  - Teva Investigational Site 11532, St Louis, Missouri
  - Teva Investigational Site 10518, Bellevue, Nebraska
  - Teva Investigational Site 10550, Omaha, Nebraska
  - Teva Investigational Site 11529, Omaha, Nebraska
  - Teva Investigational Site 11571, Las Vegas, Nevada
  - Teva Investigational Site 10559, Cherry Hill, New Jersey
  - Teva Investigational Site 11566, Edison, New Jersey
  - Teva Investigational Site 10501, Hillsborough, New Jersey
  - Teva Investigational Site 11550, Ocean City, New Jersey
  - Teva Investigational Site 10588, West Orange, New Jersey
  - Teva Investigational Site 11503, Albuquerque, New Mexico
  - Teva Investigational Site 10587, Brooklyn, New York
  - Teva Investigational Site 10520, New York, New York
  - Teva Investigational Site 10532, Newburgh, New York
  - Teva Investigational Site 10567, North Syracuse, New York
  - Teva Investigational Site 10512, Rochester, New York
  - Teva Investigational Site 10580, The Bronx, New York
  - Teva Investigational Site 10522, Canton, Ohio
  - Teva Investigational Site 10507, Cincinnati, Ohio
  - Teva Investigational Site 10523, Cincinnati, Ohio
  - Teva Investigational Site 10544, Columbus, Ohio
  - Teva Investigational Site 11521, Dayton, Ohio
  - Teva Investigational Site 11505, Middleburg Heights, Ohio
  - Teva Investigational Site 10560, Oklahoma City, Oklahoma
  - Teva Investigational Site 10574, Oklahoma City, Oklahoma
  - Teva Investigational Site 10579, Oklahoma City, Oklahoma
  - Teva Investigational Site 11544, Tulsa, Oklahoma
  - Teva Investigational Site 10598, Ashland, Oregon
  - Teva Investigational Site 11543, Medford, Oregon
  - Teva Investigational Site 11557, Portland, Oregon
  - Teva Investigational Site 10509, Altoona, Pennsylvania
  - Teva Investigational Site 10555, Philadelphia, Pennsylvania
  - Teva Investigational Site 10566, Pittsburgh, Pennsylvania
  - Teva Investigational Site 10521, Upland, Pennsylvania
  - Teva Investigational Site 10581, Lincoln, Rhode Island
  - Teva Investigational Site 10562, Providence, Rhode Island
  - Teva Investigational Site 10526, Charleston, South Carolina
  - Teva Investigational Site 11547, Charleston, South Carolina
  - Teva Investigational Site 10583, Orangeburg, South Carolina
  - Teva Investigational Site 10517, Spartanburg, South Carolina
  - Teva Investigational Site 11515, Spartanburg, South Carolina
  - Teva Investigational Site 10519, Boerne, Texas
  - Teva Investigational Site 10541, Dallas, Texas
  - Teva Investigational Site 10542, Dallas, Texas
  - Teva Investigational Site 10548, El Paso, Texas
  - Teva Investigational Site 11552, El Paso, Texas
  - Teva Investigational Site 11512, Fort Worth, Texas
  - Teva Investigational Site 11565, Houston, Texas
  - Teva Investigational Site 11568, Houston, Texas
  - Teva Investigational Site 10515, San Antonio, Texas
  - Teva Investigational Site 10569, San Antonio, Texas
  - Teva Investigational Site 11517, San Antonio, Texas
  - Teva Investigational Site 11519, San Antonio, Texas
  - Teva Investigational Site 11560, Waco, Texas
  - Teva Investigational Site 11528, Layton, Utah
  - Teva Investigational Site 10576, Provo, Utah
  - Teva Investigational Site 10534, South Burlington, Vermont
  - Teva Investigational Site 10502, Fairfax, Virginia
  - Teva Investigational Site 10595, Manassas, Virginia
  - Teva Investigational Site 10508, Richmond, Virginia
  - Teva Investigational Site 11561, Bellingham, Washington
  - Teva Investigational Site 11541, Seattle, Washington
  - Teva Investigational Site 10524, Spokane, Washington
  - Teva Investigational Site 10530, Tacoma, Washington
  - Teva Investigational Site 11511, Tacoma, Washington
  - Teva Investigational Site 10570, Greenfield, Wisconsin
  - Teva Investigational Site 11559, Greenfield, Wisconsin
- Australia (2):
  - Teva Investigational Site 85570, Bedford Park
  - Teva Investigational Site 85571, Parkville
- Bulgaria (9):
  - Teva Investigational Site 59507, Burgas
  - Teva Investigational Site 59503, Lovech
  - Teva Investigational Site 59506, Pleven
  - Teva Investigational Site 59504, Rousse
  - Teva Investigational Site 59501, Sofia
  - Teva Investigational Site 59502, Sofia
  - Teva Investigational Site 59505, Sofia
  - Teva Investigational Site 59508, Sofia
  - Teva Investigational Site 59509, Varna
- Canada (5):
  - Teva Investigational Site 11594, Burlington, Ontario
  - Teva Investigational Site 11595, Etobicoke, Ontario
  - Teva Investigational Site 11592, Sarnia, Ontario
  - Teva Investigational Site 11590, Toronto, Ontario
  - Teva Investigational Site 11591, Newmarket
- Croatia (4):
  - Teva Investigational Site 85501, Zagreb
  - Teva Investigational Site 85502, Zagreb
  - Teva Investigational Site 85503, Zagreb
  - Teva Investigational Site 85504, Zagreb
- Germany (15):
  - Teva Investigational Site 70561, Berlin
  - Teva Investigational Site 70564, Bonn
  - Teva Investigational Site 70557, Cottbus
  - Teva Investigational Site 70553, Delitzsch
  - Teva Investigational Site 70558, Frankfurt
  - Teva Investigational Site 70562, Hamburg
  - Teva Investigational Site 70560, Hanover
  - Teva Investigational Site 70555, Leipzig
  - Teva Investigational Site 70556, Magdeburg
  - Teva Investigational Site 70550, München
  - Teva Investigational Site 70554, München
  - Teva Investigational Site 70552, Münster
  - Teva Investigational Site 70563, Nuremberg
  - Teva Investigational Site 70551, Rüdersdorf
  - Teva Investigational Site 70559, Wiesbaden
- Greece (5):
  - Teva Investigational Site 85533, Athens
  - Teva Investigational Site 85534, Athens
  - Teva Investigational Site 85531, Heraklion
  - Teva Investigational Site 85532, Larissa
  - Teva Investigational Site 85530, Thessaloniki
- Hungary (16):
  - Teva Investigational Site 36507, Balassagyarmat
  - Teva Investigational Site 36504, Budapest
  - Teva Investigational Site 36505, Budapest
  - Teva Investigational Site 36514, Csoma
  - Teva Investigational Site 36516, Érd
  - Teva Investigational Site 36513, Kaba
  - Teva Investigational Site 36515, Kaposvár
  - Teva Investigational Site 36503, Miskolc
  - Teva Investigational Site 36502, Nyíregyháza
  - Teva Investigational Site 36510, Siófok
  - Teva Investigational Site 36517, Szarvas
  - Teva Investigational Site 36508, Százhalombatta
  - Teva Investigational Site 36506, Szeged
  - Teva Investigational Site 36509, Szeged
  - Teva Investigational Site 36501, Szombathely
  - Teva Investigational Site 36512, Veszprém
- Ireland (2):
  - Teva Investigational Site 59550, Dublin
  - Teva Investigational Site 59551, Dublin
- Israel (12):
  - Teva Investigational Site 72511, Ashkelon
  - Teva Investigational Site 72501, Haifa
  - Teva Investigational Site 72512, Haifa
  - Teva Investigational Site 72502, Jerusalem
  - Teva Investigational Site 72504, Jerusalem
  - Teva Investigational Site 72509, Kfar Saba
  - Teva Investigational Site 72506, Petah Tikva
  - Teva Investigational Site 72507, Ramat Gan
  - Teva Investigational Site 72503, Rehovot
  - Teva Investigational Site 72508, Tel Aviv
  - Teva Investigational Site 72510, Tel Aviv
  - Teva Investigational Site 72505, Ẕerifin
- New Zealand (4):
  - Teva Investigational Site 81571, Auckland
  - Teva Investigational Site 81572, Christchurch
  - Teva Investigational Site 81573, Tauranga
  - Teva Investigational Site 81570, Wellington
- Poland (11):
  - Teva Investigational Site 48507, Bialystok
  - Teva Investigational Site 48505, Bydgoszcz
  - Teva Investigational Site 48506, Grodzisk Mazowiecki
  - Teva Investigational Site 48501, Lodz
  - Teva Investigational Site 48509, Lodz
  - Teva Investigational Site 48513, Lublin
  - Teva Investigational Site 48508, Poznan
  - Teva Investigational Site 48512, Poznan
  - Teva Investigational Site 48502, Strzelce Opolskie
  - Teva Investigational Site 48503, Tarnów
  - Teva Investigational Site 48504, Wroclaw
- Romania (10):
  - Teva Investigational Site 81534, Brasov
  - Teva Investigational Site 81539, Brasov
  - Teva Investigational Site 81533, Bucharest
  - Teva Investigational Site 81535, Bucharest
  - Teva Investigational Site 81537, Bucharest
  - Teva Investigational Site 81531, Cluj-Napoca
  - Teva Investigational Site 81536, Cluj-Napoca
  - Teva Investigational Site 81530, Târgu Mureş
  - Teva Investigational Site 81532, Timișoara
  - Teva Investigational Site 81538, Timișoara
- Russia (12):
  - Teva Investigational Site 70505, Barnaul
  - Teva Investigational Site 70502, Kazan'
  - Teva Investigational Site 70511, Moscow
  - Teva Investigational Site 70512, Moscow
  - Teva Investigational Site 70508, Ryazan
  - Teva Investigational Site 70501, Saint Petersburg
  - Teva Investigational Site 70504, Saint Petersburg
  - Teva Investigational Site 70510, Saint Petersburg
  - Teva Investigational Site 70509, Samara
  - Teva Investigational Site 70507, Smolensk
  - Teva Investigational Site 70506, Tomsk
  - Teva Investigational Site 70503, Yaroslavl
- Teva Investigational Site 81501, Belgrade, Serbia
- South Africa (6):
  - Teva Investigational Site 36551, Bloemfontein
  - Teva Investigational Site 36552, Cape Town
  - Teva Investigational Site 36555, Cape Town
  - Teva Investigational Site 36550, Port Elizabeth
  - Teva Investigational Site 36553, Thabazimbi
  - Teva Investigational Site 36554, Witbank
- Spain (11):
  - Teva Investigational Site 34507, Aranjuez
  - Teva Investigational Site 34501, Badalona
  - Teva Investigational Site 34502, Barcelona
  - Teva Investigational Site 34510, Barcelona
  - Teva Investigational Site 34509, Bilbao
  - Teva Investigational Site 34506, Lleida
  - Teva Investigational Site 34505, Madrid
  - Teva Investigational Site 34503, Salt
  - Teva Investigational Site 34504, Santiago de Compostela
  - Teva Investigational Site 34508, Valencia
  - Teva Investigational Site 34511, Vitoria-Gasteiz
- Ukraine (22):
  - Teva Investigational Site 80501, Dnipropetrovsk
  - Teva Investigational Site 80513, Dnipropetrovsk
  - Teva Investigational Site 80511, Donetsk
  - Teva Investigational Site 80502, Kharkiv
  - Teva Investigational Site 80503, Kharkiv
  - Teva Investigational Site 80504, Kyiv
  - Teva Investigational Site 80505, Kyiv
  - Teva Investigational Site 80506, Kyiv
  - Teva Investigational Site 80507, Kyiv
  - Teva Investigational Site 80508, Kyiv
  - Teva Investigational Site 80509, Kyiv
  - Teva Investigational Site 80517, Kyiv
  - Teva Investigational Site 80519, Kyiv
  - Teva Investigational Site 80520, Kyiv
  - Teva Investigational Site 80521, Kyiv
  - Teva Investigational Site 80514, Odesa
  - Teva Investigational Site 80516, Simferopol
  - Teva Investigational Site 80512, Vinnytsia
  - Teva Investigational Site 80515, Yalta
  - Teva Investigational Site 80522, Zaporizhia
  - Teva Investigational Site 80510, Zaporizhzhia
  - Teva Investigational Site 80518, Zaporizhzhya
- United Kingdom (5):
  - Teva Investigational Site 34582, Cottingham
  - Teva Investigational Site 34584, London
  - Teva Investigational Site 34585, Penzance
  - Teva Investigational Site 34580, Torpoint
  - Teva Investigational Site 34581, Watford

REFERENCES:
- [Derived] Bernstein DI, Gillespie M, Song S, Steinfeld J. Safety, efficacy, and dose response of fluticasone propionate delivered via the novel MDPI in patients with severe asthma: A randomized, controlled, dose-ranging study. J Asthma. 2017 Aug;54(6):559-569. doi: 10.1080/02770903.2016.1242137. Epub 2016 Oct 24. PMID 27937064

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1238 subjects with asthma at 180 centers were screened for enrollment. 889 subjects met entry criteria and were enrolled into the run-in period of the study. Of the 349 subjects who were not enrolled, 337 were excluded on the basis of inclusion/exclusion criteria, 5 subjects withdrew consent, and for 6 the reason given was "other".
Groups:
- Placebo MDPI (Run-In): Upon enrollment, participants used current asthma medications and 1 inhalation of placebo multidose dry powder inhaler (MDPI), single-blind, twice daily for 14-day (±2 days).
Period: Pre-Assignment Period (Run-In Placebo)
Arm/Group | Placebo MDPI (Run-In) | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Started | 889 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 640 (Participants randomized into the Treatment Period) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 249 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Inclusion/exclusion criteria | 49 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomization criteria not met | 166 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 15 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Placebo MDPI (Run-In) | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Started | 0 | 107 | 107 | 106 | 107 | 106 | 107
Safety Population | 0 | 107 | 107 | 106 | 107 | 106 | 106
Efficacy Population (Full Analysis Set) | 0 | 107 | 106 | 102 | 107 | 105 | 103
Completed | 0 | 82 | 87 | 75 | 80 | 58 | 77
Not Completed | 0 | 25 | 20 | 31 | 27 | 48 | 30
Not completed — Adverse Event | 0 | 1 | 1 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 2 | 4 | 2
Not completed — Physician Decision | 0 | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 5 | 4 | 10 | 6 | 8 | 12
Not completed — Sponsor request | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Met stopping criteria | 0 | 16 | 13 | 19 | 16 | 33 | 15
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Noncompliance to study medication | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg | Total
Number analyzed (Participants) | 107 | 107 | 106 | 107 | 106 | 107 | 640
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (14.59) | 48.7 (12.48) | 47.7 (14.18) | 50.9 (13.32) | 49.8 (12.87) | 49.2 (13.26) | 49.0 (13.46)
Age, Customized [Number; unit: participants]
  Adolescents (12-17 years) | 2 | 3 | 1 | 1 | 1 | 1 | 9
  Adults (18-64 years) | 94 | 99 | 90 | 90 | 94 | 96 | 563
  Adults (65-84 years) | 11 | 5 | 15 | 16 | 11 | 10 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 55 | 66 | 72 | 65 | 58 | 379
  Male | 44 | 52 | 40 | 35 | 41 | 49 | 261
Race/Ethnicity, Customized [Number; unit: participants]
  White | 96 | 94 | 93 | 91 | 96 | 95 | 565
  Black | 9 | 12 | 12 | 13 | 8 | 11 | 65
  Asian | 1 | 1 | 1 | 2 | 2 | 0 | 7
  American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 5 | 7 | 8 | 12 | 6 | 9 | 47
  Not Hispanic or Latino | 102 | 100 | 98 | 95 | 100 | 98 | 593
Weight [Mean (Standard Deviation); unit: kg] | 86.7 (23.73) | 86.6 (22.90) | 84.4 (21.89) | 84.4 (20.56) | 86.2 (25.19) | 83.3 (16.76) | 85.3 (21.95)
Height [Mean (Standard Deviation); unit: cm] | 169.4 (13.04) | 168.7 (9.14) | 168.4 (7.86) | 167.4 (9.67) | 168.1 (8.57) | 168.0 (8.33) | 168.3 (9.58)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.3 (17.88) | 30.4 (7.60) | 29.8 (8.12) | 30.1 (6.81) | 30.5 (8.83) | 29.6 (6.03) | 30.3 (10.02)
Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] | 2.108 (0.662) | 2.031 (0.551) | 1.999 (0.525) | 2.016 (0.636) | 1.984 (0.565) | 1.955 (0.529) | 2.016 (0.579)
% Predicted Expiratory Volume In 1 Second [Mean (Standard Deviation); unit: percent predicted FEV1] | 63.7 (10.9) | 63.1 (9.5) | 63.4 (12.1) | 65.3 (11.4) | 63.1 (10.0) | 62.5 (12.1) | 63.5 (11.0)
Qualifying Airway Reversibility [Mean (Standard Deviation); unit: percentage increase in FEV1] — Patients demonstrated a ≥12% reversibility of FEV1 within 30 minutes following 2-4 inhalations of albuterol/salbutamol inhalation aerosol at the screening visit. If subjects failed to demonstrate an increase in FEV1 ≥12% then subjects were not eligible for the study; however, based on investigator judgment, they were allowed to retest once within 7 days. Reversibility values of 11.50 through 11.99% were rounded to 12%. Documented historical reversibility of ≥12 % within 1 year was accepted.
  percentage increase in FEV1 | 31.6 (22.4) | 27.3 (14.7) | 30.4 (25.2) | 29.1 (19.5) | 28.9 (19.1) | 26.8 (15.7) | 29.0 (19.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Trough (Morning Predose And Pre-Rescue Bronchodilator) Forced Expiratory Volume In 1 Second (FEV1) Over The 12-Week Treatment Period
Description: Trough FEV1 was measured electronically by spirometry at morning (AM) investigational site visits, before administration of the AM dose of study drug, and before albuterol/salbutamol administration. The highest FEV1 value from 3 acceptable and 2 reproducible maneuvers was used. All FEV1 data were submitted to a central reading center for evaluation.
  The p-values for the treatment comparisons to placebo are from an MMRM model excluding FLOVENT DISKUS data: change from baseline = baseline FEV1 + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Day 1 pre-dose), Weeks 1, 2, 3, 4, 6, 8, 10 and 12
Population: Full analysis set, including participants who contributed at least once to the analysis. Based on blinded data review, data from one site are excluded due to good clinical practice (GCP) concerns. Flovent Diskus data was used for confirmatory and exploratory endpoints; FEV1 data for Flovent Diskus is reported in outcome #12.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 104 | 102 | 97 | 103 | 98 | 0
liters | 0.059 (0.0269) | 0.101 (0.0268) | 0.109 (0.0278) | 0.125 (0.0274) | 0.053 (0.0283) |
Statistical Analysis 1: Comparison: Fp MDPI 50 mcg vs Fp MDPI 100 mcg vs Fp MDPI 200 mcg vs Fp MDPI 400 mcg vs Placebo MDPI; A linear in log-dose trend contrast was constructed to evaluate the time-averaged dose-response trend, where the logarithm of dose was defined as log(dose+1) to accommodate the case of a zero dose (placebo). A fixed-sequence testing procedure was employed to control the overall Type I error rate at the 0.05 level. Specifically, the 2-sided linear in log-dose time-averaged trend test was first performed at the 0.05 level of significance; Test type: Superiority or Other; p = 0.0604, Regression, Linear — If the Fp MDPI showed a significantly positive trend, then contrasts for pairwise comparisons of each Fp MDPI dose versus placebo were done in the sequence of highest to lowest Fp MDPI dose
Statistical Analysis 2: Comparison: Fp MDPI 400 mcg vs Placebo MDPI; No explicit structure was assumed for the covariance among the repeated measures. Analyses for comparison of Fp MDPI to placebo did not contain FLOVENT DISKUS data; Test type: Superiority or Other; p = 0.0637, mixed model for repeated measures — Significance at the 0.05 level; LSM difference = 0.072, 95% CI 2-sided [-0.004 to 0.149] — Fp 400 - Placebo
Statistical Analysis 3: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1585, mixed model for repeated measures — Significance at the 0.05 level; LSM difference = 0.056, 95% CI 2-sided [-0.022 to 0.133] — Fp 200 - Placebo
Statistical Analysis 4: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2221, mixed model for repeated measures — Significance at the 0.05 level; LSM difference = 0.048, 95% CI 2-sided [-0.029 to 0.124] — Fp 100 - Placebo
Statistical Analysis 5: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8694, mixed model for repeated measures — Significance at the 0.05 level; LSM difference = 0.006, 95% CI 2-sided [-0.070 to 0.083] — Fp 50 - Placebo

2. Secondary Outcome: Change From Baseline In Weekly Average Of Daily Trough (Predose And Pre-Rescue Bronchodilator) Morning Peak Expiratory Flow (PEF) Over The 12-Week Treatment Period
Description: Peak expiratory flow was determined in the AM and in the PM, before administration of study or rescue medications using a handheld electronic peak flow meter. The highest value of triplicate measurements obtained was recorded by the subject's diary device.
  On mornings for which a treatment visit was scheduled (TV1 through TV9), the PEF was measured and recorded at the investigational site visit.
  Baseline trough AM PEF was defined as the average of recorded (non-missing) trough AM PEF assessments over the 7 days directly preceding first study drug intake.
  The p-values for the treatment comparisons to placebo are from an MMRM model excluding FLOVENT DISKUS data: change from baseline = baseline PEF + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Days -6 to Day 1 pre-dose), Weeks 1, 2, 3, 4, 6, 8, 10 and 12
Population: Full analysis set, including participants who contributed at least once to the analysis. Based on blinded data review, data from one site are excluded due to good clinical practice (GCP) concerns. Flovent Diskus data was used for confirmatory and exploratory endpoints; morning PEF data for Flovent Diskus is reported in outcome #13.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 101 | 101 | 96 | 101 | 98 | 0
liters/minute | 10.48 (4.299) | 9.34 (4.245) | 10.03 (4.420) | 9.61 (4.307) | 2.24 (4.507) |
Statistical Analysis 1: Comparison: Fp MDPI 50 mcg vs Fp MDPI 100 mcg vs Fp MDPI 200 mcg vs Fp MDPI 400 mcg vs Placebo MDPI vs Flovent Diskus 250mcg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1512, Regression, Linear — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fp MDPI 400 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2361, Regression, Linear — Significance at the 0.05 level; LSM difference = 7.36, 95% CI 2-sided [-4.83 to 19.56]
Statistical Analysis 3: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2169, Regression, Linear; Significance at the 0.05 level; LSM difference = 7.78, 95% CI 2-sided [-4.59 to 20.15]
Statistical Analysis 4: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2523, Regression, Linear — Significance at the 0.05 level; LSM difference = 7.09, 95% CI 2-sided [-5.07 to 19.26]
Statistical Analysis 5: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1858, Regression, Linear — Significance at the 0.05 level; LSM difference = 8.23, 95% CI 2-sided [-3.98 to 20.45]

3. Secondary Outcome: Change From Baseline In Weekly Average Of Daily Trough (Predose And Pre-Rescue Bronchodilator) Evening Peak Expiratory Flow (PEF) Over The 12-Week Treatment Period
Description: Peak expiratory flow was determined in the AM and in the PM, before administration of study or rescue medications using a handheld electronic peak flow meter. The highest value of triplicate measurements obtained was recorded by the subject's diary device.
  PM PEF baseline was defined as the average of recorded (nonmissing) PM PEF assessments over the 7 days directly preceding first study drug intake.
  The p-values for the treatment comparisons to placebo are from an MMRM model excluding FLOVENT DISKUS data: change from baseline = baseline PEF + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Days -6 to Day 1 pre-dose), Weeks 1, 2, 3, 4, 6, 8, 10 and 12
Population: Full analysis set, including participants who contributed at least once to the analysis. Based on blinded data review, data from one site are excluded due to good clinical practice (GCP) concerns. Flovent Diskus data was used for confirmatory and exploratory endpoints; evening PEF data for Flovent Diskus is reported in outcome #14.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 103 | 99 | 96 | 102 | 96 | 0
liters/minute | 3.81 (4.183) | 6.41 (4.209) | 7.45 (4.335) | 10.97 (4.208) | 3.42 (4.462) |
Statistical Analysis 1: Comparison: Fp MDPI 50 mcg vs Fp MDPI 100 mcg vs Fp MDPI 200 mcg vs Fp MDPI 400 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2879, Regression, Linear — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fp MDPI 400 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2166, Regression, Linear — Significance at the 0.05 level; LSM difference = 7.56, 95% CI 2-sided [-4.45 to 19.56]
Statistical Analysis 3: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5167, Regression, Linear — Significance at the 0.05 level; LSM difference = 4.03, 95% CI 2-sided [-8.17 to 16.23]
Statistical Analysis 4: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6258, Regression, Linear — Significance at the 0.05 level; LSM difference = 2.99, 95% CI 2-sided [-9.06 to 15.05]
Statistical Analysis 5: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9487, Regression, Linear — Significance at the 0.05 level; LSM difference = 0.39, 95% CI 2-sided [-11.60 to 12.39]

4. Secondary Outcome: The Kaplan-Meier Estimate Of The Probability Of Remaining In The Study At Week 12
Description: The analysis of probability of remaining in the study at Week 12 used the time to patient withdrawal for worsening asthma. Worsening asthma was defined as:
  1. clinic visit FEV1 below the FEV1 stability limit value calculated on Day 1.
  2. any 7-day run-in or treatment window (using information from the patient diary) during which the subject experienced:
     * 3 or more days in which the highest PEF has fallen below the PEF stability limit calculated on Day 1
     * 3 or more days in which ≥12 inhalations/day of albuterol/salbutamol was used
     * 2 or more days in which the subject experienced a nighttime asthma symptom score of >2
  3. clinical asthma exacerbation, defined as worsening asthma requiring any treatment other than study drug or rescue albuterol/salbutamol including the use of systemic corticosteroids and/or ER visit or hospitalization.
  Patients who had withdrawn due to reasons other than worsening asthma were right-censored at the date of last assessment.
Time Frame: Day 1 to Week 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 107 | 106 | 102 | 107 | 105 | 103
probability | 0.6872 [0.5891 to 0.7665] | 0.6330 [0.5307 to 0.7188] | 0.5852 [0.4796 to 0.6766] | 0.6109 [0.5093 to 0.6977] | 0.4722 [0.3712 to 0.5665] | 0.5657 [0.4617 to 0.6571]
Statistical Analysis 1: Comparison: Fp MDPI 400 mcg vs Placebo MDPI; P-value for comparison of survival curve to placebo; Test type: Superiority or Other; p = 0.0341, Log Rank — Significance level of 0.05
Statistical Analysis 2: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; P-value for comparison of survival curve to placebo; Test type: Superiority or Other; p = 0.0340, Log Rank — Significance level of 0.05
Statistical Analysis 3: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; P-value for comparison of survival curve to placebo; Test type: Superiority or Other; p = 0.0058, Log Rank — Significance level of 0.05
Statistical Analysis 4: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; P-value for comparison of survival curve to placebo; Test type: Superiority or Other; p = 0.0018, Log Rank — Significance level of 0.05
Statistical Analysis 5: Comparison: Placebo MDPI vs Flovent Diskus 250mcg; P-value for comparison of survival curve to placebo; Test type: Superiority or Other; p = 0.1006, Log Rank — Significance level of 0.05

5. Secondary Outcome: Change From Baseline In The Percentage Of Rescue-Free 24-Hour Periods
Description: The change from baseline in the percentage of rescue-free 24-hour periods was analyzed with a marginal (also called population averaged) logistic model, with the response being the proportion of rescue-free 24-hour periods. The model included 2 time points of measurement for each subject: the baseline (the last 7 days before the treatment period) and the treatment period. The model contained covariates for sex, age, and treatment. Rescue-free days were as indicated in patient diaries.
  Data values are estimated means.
Time Frame: Baseline (Day -6 to Day 1 predose), Treatment (Day 1 to Week 12)
Population: Full analysis set including participants who contributed at least once to the analysis.
Measure: Mean (Standard Error); unit: percentage of total 24 hour periods
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 96 | 90 | 91 | 99 | 93 | 95
percentage of total 24 hour periods | 22.78 (4.016) | 26.41 (4.013) | 16.18 (3.662) | 28.05 (3.951) | 27.15 (4.475) | 15.87 (3.750)
Statistical Analysis 1: Comparison: Fp MDPI 400 mcg vs Placebo MDPI; Estimates computed from a generalized linear logistic model with gender and age as covariates and allows correlation between estimates on the same subject. Interpretation of the estimates is that they are the average over the population at the average level of continuous covariate (age) averaged over discrete covariate (gender); Test type: Superiority or Other; p = 0.88116, Regression, Linear — Significance at the 0.05 level; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [-11.12 to 12.91]
Statistical Analysis 2: Comparison: Fp MDPI 200 mcg vs Placebo MDPI; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.05977, Regression, Linear — Significance at the 0.05 level; Mean Difference (Final Values) = -10.98, 95% CI 2-sided [-22.64 to 0.68]
Statistical Analysis 3: Comparison: Fp MDPI 100 mcg vs Placebo MDPI; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.90426, Regression, Linear — Significance at the 0.05 level; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-13.02 to 11.54]
Statistical Analysis 4: Comparison: Fp MDPI 50 mcg vs Placebo MDPI; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.47310, Regression, Linear — Significance at the 0.05 level; Mean Difference (Final Values) = -4.38, 95% CI 2-sided [-16.57 to 7.82]

6. Secondary Outcome: Area Under The Plasma Concentration-Time Curve From Time Zero To The Time Of The Last Measurable Concentration (AUC0-t)
Time Frame: Day 1 predose (within 10 minutes of treatment administration), and 5, 10, 15, 30, and 45 minutes, 1 hour, 1 hour 15 minutes, 1 hour 30 minutes, and 2, 4, 8, and 12 hours postdose
Population: Pharmacokinetic analysis set. Two participants in the Fp MDPI 100 mcg treatment arm did not have AUC data. PK tests not run on participants in the Placebo MDPI arm.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 18 | 16 | 18 | 20 | 0 | 16
pg*hr/mL | 117.6 (145.79) | 126.8 (33.73) | 292.0 (162.28) | 462.8 (262.45) |  | 162.3 (74.79)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 18 | 16 | 18 | 20 | 0 | 16
pg/mL | 19.1 (15.53) | 26.5 (6.16) | 55.2 (29.12) | 83.0 (44.32) |  | 32.5 (13.92)

8. Secondary Outcome: Time Of Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 18 | 16 | 18 | 20 | 0 | 16
hours | 1.0 (0.54) | 1.2 (1.85) | 2.2 (3.58) | 1.4 (2.60) |  | 1.8 (2.75)

9. Secondary Outcome: Patients With Treatment-Emergent Adverse Experiences (TEAE) During the Treatment Period
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Week 12
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 107 | 107 | 106 | 107 | 106 | 106
participants
  Any adverse event (AE) | 31 | 27 | 34 | 41 | 33 | 27
  Severe AE | 3 | 1 | 1 | 1 | 1 | 0
  Treatment-related AE | 4 | 1 | 6 | 9 | 5 | 2
  Deaths | 0 | 0 | 0 | 0 | 0 | 0
  Other serious AEs | 1 | 1 | 1 | 0 | 1 | 0
  Withdrawn from treatment due to AEs | 1 | 1 | 1 | 1 | 1 | 0

10. Secondary Outcome: Patients With Positive Swab Test Results for Oral Candidiasis
Description: Oropharyngeal examinations for visual evidence of oral candidiasis were conducted at each visit. Any visual evidence of oral candidiasis during the oropharyngeal exam was evaluated by obtaining and analyzing a swab of the suspect area.
  This outcomes indicates how many patients had positive swab test results. The total number of patients who had oropharyngeal exams at each timepoint are specified in the timepoint field. Appropriate therapy was to be initiated immediately at the discretion of the investigator and was not to be delayed for culture confirmation. Subjects with a culture-positive infection could continue participation in the study on appropriate anti-infective therapy, provided this therapy was not prohibited by the protocol.
Time Frame: Screening (Days -21 to -14), Randomization (Day 1), Weeks 1, 2, 3, 4, 6, 8, 10, 12
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 107 | 107 | 106 | 107 | 106 | 106
participants
  Screening: number analyzed (Participants) | 107 | 106 | 106 | 107 | 106 | 104
  Screening | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 | 0 | 0 | 1 | 0 | 1 | 1
  Week 1: number analyzed (Participants) | 102 | 103 | 98 | 97 | 96 | 99
  Week 1 | 0 | 0 | 0 | 0 | 1 | 1
  Week 2: number analyzed (Participants) | 99 | 101 | 94 | 95 | 84 | 92
  Week 2 | 0 | 0 | 1 | 2 | 0 | 0
  Week 3: number analyzed (Participants) | 91 | 98 | 92 | 93 | 80 | 87
  Week 3 | 0 | 0 | 0 | 4 | 0 | 0
  Week 4: number analyzed (Participants) | 91 | 95 | 88 | 87 | 75 | 87
  Week 4 | 1 | 0 | 1 | 1 | 0 | 0
  Week 6: number analyzed (Participants) | 86 | 92 | 86 | 86 | 68 | 85
  Week 6 | 0 | 0 | 0 | 1 | 0 | 0
  Week 8: number analyzed (Participants) | 83 | 90 | 81 | 83 | 64 | 82
  Week 8 | 0 | 0 | 1 | 0 | 0 | 1
  Week 10: number analyzed (Participants) | 83 | 87 | 77 | 82 | 60 | 79
  Week 10 | 0 | 0 | 0 | 1 | 0 | 0
  Week 12: number analyzed (Participants) | 104 | 104 | 103 | 106 | 102 | 100
  Week 12 | 0 | 0 | 0 | 1 | 0 | 1

11. Secondary Outcome: 24-Hour Urinary Cortisol Excretion at Baseline, Week 12 and Endpoint
Description: 24-hour urinary cortisol excretion was determined from 24-hour pooled-urine samples; urine was refrigerated until return to the investigational site after each 24-hour collection period. Urine was collected within 7 days of Day 1 and within 7 days of Week 12. Urine cortisol sample collection was not required at endpoint visit for subjects who terminated early from the study.
Time Frame: Baseline (Day 1), Week 12, Endpoint
Population: Urine cortisol analysis set
Measure: Mean (Standard Deviation); unit: nmol/day
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 62 | 70 | 55 | 68 | 41 | 59
nmol/day
  Baseline | 65.3 (42.69) | 63.8 (44.70) | 66.6 (45.53) | 57.4 (34.68) | 74.3 (43.54) | 66.2 (42.68)
  Week 12: number analyzed (Participants) | 61 | 70 | 53 | 65 | 38 | 57
  Week 12 | 71.8 (48.37) | 61.5 (45.73) | 66.8 (53.96) | 46.2 (38.67) | 69.2 (49.56) | 58.5 (43.75)
  Endpoint | 71.0 (48.31) | 61.5 (45.73) | 65.8 (53.33) | 45.0 (38.33) | 74.4 (54.97) | 58.4 (43.49)

12. Other Pre Specified Outcome: Change From Baseline In Trough (Morning Predose And Pre-Rescue Bronchodilator) Forced Expiratory Volume In 1 Second (FEV1) Over The 12-Week Treatment Period (Including the Flovent Diskus Treatment Arm)
Description: Peak expiratory flow was determined in the AM and in the PM, before administration of study or rescue medications using a handheld electronic peak flow meter. The highest value of triplicate measurements obtained was recorded by the subject's diary device.
  On mornings for which a treatment visit was scheduled (TV1 through TV9), the PEF was measured and recorded at the investigational site visit.
  Baseline trough AM PEF was defined as the average of recorded (nonmissing) trough AM PEF assessments over the 7 days directly preceding first study drug intake.
  The p-values for the treatment comparisons to Flovent Diskus are from an MMRM model which includes data from all treatments: change from baseline = baseline PEF + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Day 1 pre-dose), Weeks 1, 2, 3, 4, 6, 8, 10 and 12
Population: Full analysis set, including participants who contributed at least once to the analysis. Based on blinded data review, data from one site are excluded due to good clinical practice (GCP) concerns.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 104 | 102 | 97 | 103 | 98 | 100
liters | 0.063 (0.027) | 0.102 (0.0269) | 0.113 (0.0279) | 0.129 (0.0274) | 0.057 (0.0284) | 0.110 (0.0274)
Statistical Analysis 1: Comparison: Fp MDPI 400 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.6161, mixed model for repeated measures — 0.05 level of significance; LSM difference = 0.019, 95% CI 2-sided [-0.057 to 0.096]
Statistical Analysis 2: Comparison: Fp MDPI 200 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.9245, mixed model for repeated measures — 0.05 level of significance; LSM difference = 0.004, 95% CI 2-sided [-0.973 to 0.080]
Statistical Analysis 3: Comparison: Fp MDPI 100 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.8434, mixed model for repeated measures — 0.05 level of significance; LSM difference = -0.008, 95% CI 2-sided [-0.083 to 0.068]
Statistical Analysis 4: Comparison: Fp MDPI 50 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.2241, mixed model for repeated measures — 0.05 level of significance; LSM difference = -0.047, 95% CI 2-sided [-0.122 to 0.029]
Statistical Analysis 5: Comparison: Placebo MDPI vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.1822, mixed model for repeated measures — 0.05 level of significance; LSM difference = -0.053, 95% CI 2-sided [-0.130 to 0.025]

13. Other Pre Specified Outcome: Change From Baseline In Weekly Average Of Daily Trough (Predose And Pre-Rescue Bronchodilator) Morning Peak Expiratory Flow (PEF) Over The 12-Week Treatment Period (Including the Flovent Diskus Treatment Arm)
Description: Peak expiratory flow was determined in the AM and in the PM, before administration of study or rescue medications using a handheld electronic peak flow meter. The highest value of triplicate measurements obtained was recorded by the subject's diary device.
  On mornings for which a treatment visit was scheduled (TV1 through TV9), the PEF was measured and recorded at the investigational site visit.
  Baseline trough AM PEF was defined as the average of recorded (nonmissing) trough AM PEF assessments over the 7 days directly preceding first study drug intake.
  The p-values for the treatment comparisons to Flovent Diskus are from an MMRM model that included data for all treatments: change from baseline = baseline PEF + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Days -6 to Day 1 pre-dose), Weeks 1, 2, 3, 4, 6, 8, 10 and 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 101 | 101 | 96 | 101 | 98 | 99
liters/minute | 10.85 (4.245) | 9.39 (4.193) | 10.29 (4.362) | 10.40 (4.254) | 2.52 (4.453) | 15.97 (4.283)
Statistical Analysis 1: Comparison: Fp MDPI 400 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.3568, Regression, Linear — 0.05 level of significance; LSM difference = -5.56, 95% CI 2-sided [-17.42 to 6.29]
Statistical Analysis 2: Comparison: Fp MDPI 200 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.3531, Regression, Linear — 0.05 level of significance; LSM difference = -5.68, 95% CI 2-sided [-17.67 to 6.32]
Statistical Analysis 3: Comparison: Fp MDPI 100 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.2724, Regression, Linear — 0.05 level of significance; LSM difference = -6.58, 95% CI 2-sided [-18.35 to 5.19]
Statistical Analysis 4: Comparison: Fp MDPI 50 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.3964, Regression, Linear — 0.05 level of significance; LSM difference = -5.11, 95% CI 2-sided [-16.95 to 6.72]
Statistical Analysis 5: Comparison: Placebo MDPI vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.0296, Regression, Linear — 0.05 level of significance; LSM difference = -13.45, 95% CI 2-sided [-25.57 to -1.33]

14. Other Pre Specified Outcome: Change From Baseline In Weekly Average Of Daily Trough (Predose And Pre-Rescue Bronchodilator) Evening Peak Expiratory Flow (PEF) Over The 12-Week Treatment Period (Including the Flovent Diskus Treatment Arm)
Description: Peak expiratory flow was determined in the AM and in the PM, before administration of study or rescue medications using a handheld electronic peak flow meter. The highest value of triplicate measurements obtained was recorded by the subject's diary device.
  PM PEF baseline was defined as the average of recorded (nonmissing) PM PEF assessments over the 7 days directly preceding first study drug intake.
  The p-values for the treatment comparisons to Flovent Diskus are from an MMRM model that included data for all treatments: change from baseline = baseline PEF + sex + age + treatment + visit + treatment*visit with an unstructured covariance matrix assumed.
Time Frame: Baseline (Days -6 to Day 1 pre-dose), Weeks 1, 2, 3, 4, 6, 8, 10 and 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Fp MDPI 50 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Placebo MDPI | Flovent Diskus 250mcg
Number analyzed (Participants) | 103 | 99 | 96 | 102 | 96 | 99
liters/minute | 4.22 (4.245) | 6.52 (4.275) | 7.89 (4.397) | 11.72 (4.271) | 3.35 (4.518) | 12.4 (4.309)
Statistical Analysis 1: Comparison: Fp MDPI 400 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.9101, Regression, Linear — 0.05 level of significance; LSM difference = -0.69, 95% CI 2-sided [-12.59 to 11.22]
Statistical Analysis 2: Comparison: Fp MDPI 200 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.4634, Regression, Linear — 0.05 level of significance; LSM difference = -4.51, 95% CI 2-sided [-16.6 to 7.57]
Statistical Analysis 3: Comparison: Fp MDPI 100 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.3333, Regression, Linear — 0.05 level of significance; LSM difference = -5.88, 95% CI 2-sided [-17.8 to 6.05]
Statistical Analysis 4: Comparison: Fp MDPI 50 mcg vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.1763, Regression, Linear — 0.05 level of significance; LSM difference = -8.19, 95% CI 2-sided [-20.06 to 3.69]
Statistical Analysis 5: Comparison: Placebo MDPI vs Flovent Diskus 250mcg; Test type: Superiority or Other; p = 0.1469, Regression, Linear — 0.05 level of significance; Slope = -9.05, 95% CI 2-sided [-21.3 to 3.19]

ADVERSE EVENTS:
Time Frame: Day 1 to Week 16
Groups:
- Flovent Diskus 250 mcg: Fluticasone propionate (Fp) 250 mcg per dose twice a day (for a total daily dose of 500 mcg) using a multidose dry powder inhaler (MDPI) for 12 weeks in an open-label manner.
  During the run-in and the treatment periods, all subjects replaced their current rescue medication with albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI) (90 mcg/actuation) for use on an as needed basis for the relief of asthma symptoms.
Arm/Group | Flovent Diskus 250 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg | Fp MDPI 400 mcg | Fp MDPI 50 mcg | Placebo MDPI
Serious Adverse Events (participants affected / at risk) | 0/106 | 1/107 | 1/106 | 0/107 | 1/107 | 1/106
Other Adverse Events (participants affected / at risk) | 4/106 | 4/107 | 5/106 | 7/107 | 5/107 | 6/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flovent Diskus 250 mcg (N=106) | Fp MDPI 100 mcg (N=107) | Fp MDPI 200 mcg (N=106) | Fp MDPI 400 mcg (N=107) | Fp MDPI 50 mcg (N=107) | Placebo MDPI (N=106)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flovent Diskus 250 mcg (N=106) | Fp MDPI 100 mcg (N=107) | Fp MDPI 200 mcg (N=106) | Fp MDPI 400 mcg (N=107) | Fp MDPI 50 mcg (N=107) | Placebo MDPI (N=106)
Headache (Nervous system disorders) | 4 (4) | 4 (10) | 5 (6) | 7 (9) | 5 (5) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.